CLINICAL TRIAL: NCT04164316
Title: The Effects of Kinesio Taping on Biomechanical and Clinical Outcomes in Runners With Iliotibial Band Friction Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Pongchai Watcharakhueankhan, Principal Investigator, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-CIRB 2019/208.2510
Record Dates: First submitted 2019-11-08; First posted 2019-11-15 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Iliotibial Band Syndrome
Keywords: Kinesio Taping; Biomechanics; Iliotibial Band Friction Syndrome; Clinical Outcomes
MeSH Terms: conditions — Iliotibial Band Syndrome | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Exploratory Randomized Control Study
Masking Description: This is using Kinesio Tape which is difficult to blind the patients and clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Tape No Tension (Sham Comparator): Kinesio Tape No Tension
  Interventions: Device: Kinesio Tape
- Kinesio Tape with Tension (Active Comparator): Kinesio Tape with Tension
  Interventions: Device: Kinesio Tape

INTERVENTIONS:
Device: Kinesio Tape — Kinesio TexTM Tape which is the original elastic therapeutic adhesive tape which is a latex-free, hypoallergenic, waterproof, porous.

SUMMARY:
The aim of this study is to investigate the efficacy and effectiveness of the application of Kinesio Taping in the short-term management of ITBFS in an exploratory randomized control study in two patient groups, an experimental group receiving Kinesio Taping with tension, and a control group receiving Kinesio Taping with no tension.

DETAILED DESCRIPTION:
To determine the immediate effects of taping on the three-dimensional joint kinematics and moments of the lower limb during running in ITBFS patients, and to determine any differences between the experimental and control groups.

To determine the immediate effects of taping on muscle activity of the gluteus maximus, gluteus medius, tensor fascia lata, vastus medialis, and vastus lateralis in ITBFS patients, and to determine any differences between the experimental and control groups.

To determine if the short-term perceptions of pain, symptoms, ADL function, sport and recreation function, quality of Life, and fear of movement are changed with taping, and to determine any differences between the experimental and control groups.

To determine any perceived changes in the stability of the knee joint, comfort and benefits with taping, and to determine any differences between the experimental and control groups.

To determine if muscle strength, muscle length, and functional movement are changed with taping, and to determine any differences between the experimental and control groups.

To explore the relationship between the clinical and biomechanical outcome measures in ITBFS patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 45 years
* Regularly run a minimum of 10 kilometres a week,
* Current symptoms of ITBFS, assessed using the Noble compression test and Ober's test, and pain at lateral femoral condyle during running

Exclusion Criteria:

* History of taking any analgesic or anti-inflammatory drugs for 72 hours prior to testing.
* Previous surgery to the lower limbs,
* Skin allergy to kinesio tape,
* Signs or symptoms of other knee pathologies including; patellofemoral pain, knee joint osteoarthritis, lateral meniscus injury, common peroneal nerve injury, refer pain from lumbar spine, superior tibiofibular joint sprain, and popliteus or bicep femoris tendinitis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating scale | one week
  Numerical Pain Rating scale; pain intensity during running from 0 to10 scale where 0 = No pain and 10 = worst pain Imaginable.
Pelvis, Hip, Knee, and Ankle angle. | Immediately after the intervention
  Three-dimensional joint kinematics measurement by motion analysis capture
Hip, Knee, and Ankle Moments | Immediately after the intervention
  Three-dimensional joint kinematics measurement by motion analysis capture
Surface Electromyography Data | Immediately after the intervention
  Five Surface Electromyography electrodes were placed over the gluteus maximus (Gmax), gluteus medius (Gmed), tensor fascia latae (TFL), vastus medialis (VM), vastus lateralis (VL) muscles to measure muscle activity.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | one week
  The Knee Injury and Osteoarthritis Outcome Score's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
Tampa Scale for Kinesiophobia | one week
  The Tampa Scale for Kinesiophobia is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. A Likert scale is used and all items have four possible answer options scored from 1 (strongly disagree ) to 4 (strongly agree ).
Global Rating Of Change Scale | one week
  Global rating of change (GRC) scales are very commonly used in clinical research, particularly in the musculoskeletal area. the overall condition of your injured body part or region. Rating from -7 A very great deal worse to +7 scale (A very great deal better) from the begin intervention time until now.

CONTACTS AND LOCATIONS:
Overall Officials: Jim Richards, Professor, Study Director — University of Central Lancashire
Locations (2):
- Thailand (2):
  - Physical Therapy Center (Pinklao) Faculty of Physical Therapy, Mahidol University, Bangkok
  - Faculty of Physical Therapy, Mahidol University, Nakhon Pathom

IPD SHARING:
Plan to Share IPD: No
To be confirmed